CLINICAL TRIAL: NCT00944424
Title: GORG - 002 Randomized Phase III Trial to Determine the Effectiveness of High Dose Versus Standard Dose of Vitamin D2 (Ergocalciferol) Given With Docetaxel in Patients With Metastatic Breast Cancer
Brief Title: Phase III Trial of High Dose vs. Standard Dose Vit D2 With Docetaxel in Met Breast ca
Acronym: GORG-002
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAC # 2091-009
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: Vitamin D in patients with metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Ergocalciferols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Arm A = Docetaxel + High dose Vitamin D2
  Interventions: Drug: Docetaxel + High dose Vitamin D2
- Arm B (Active Comparator): Docetaxel + Standard dose Vitamin D2
  Interventions: Drug: Docetaxel + Standard dose Vitamin D2

INTERVENTIONS:
Drug: Docetaxel + High dose Vitamin D2 — Docetaxel + High dose Vitamin D2
  Arms: Arm A
Drug: Docetaxel + Standard dose Vitamin D2 — Docetaxel + Standard dose Vitamin D2
  Arms: Arm B

SUMMARY:
Randomized phase III trial to determine the effectiveness of High dose versus Standard dose of Vitamin D2 (Ergocalciferol) given with Docetaxel in patients with metastatic breast cancer

DETAILED DESCRIPTION:
2 Arms Randomization in patients with metastatic breast cancer.

Arm A = Docetaxel + High dose Vitamin D2

Arm B = Docetaxel + Standard dose Vitamin D2

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic adenocarcinoma of the breast.
* Gender: female.
* Age ≥18 years.
* ECOG performance status ≤ 2.(see appendix I)
* 25 (OH) Vitamin D level ≤ 100nmol/L (40ng/L).
* No more than 1 prior chemotherapy regimen not including Docetaxel or Paclitaxel for metastatic breast cancer.
* Patients progressed on Doxorubicin or epirubicin as first line for metastatic breast cancer is eligible.
* Concurrent bisphosphonate therapy allowed.
* Life expectancy more than 6 months
* At least 12 months since prior adjuvant or neo-adjuvant chemotherapy including Taxanes regimens.
* Adequate hematologic, hepatic and renal function.
* Written informed consent.

Exclusion Criteria:

* Pregnant or lactating women.
* Male breast cancer.
* Women of childbearing potential unless surgically sterile or using adequate measures of contraception.
* Metastatic inflammatory breast cancer.
* CNS metastasis.
* Leptomeningeal carcinomatosis.
* Malignant hypercalcemia.
* History of kidney stones.
* History of active primary hyperparathyroidism.
* Normal 25 (OH) Vitamin D level ≥100 nmol/L or ≥ 40 ng/L.
* Previous or concomitant malignancy of any type, except adequately treated basal cell carcinoma of the skin or in situ cervix cancer.
* Patient on any anti-Psychotic medications or Steroid therapy.
* History of malabsorption syndrome (pancreatic insufficiency, celiac disease and tropical sprue).
* Any of the following abnormal baseline hematological values:

  * ANC < 1.0 x109/L, or platelets < 100.000 x 109/L.
* Any of the following abnormal laboratory tests: total serum bilirubin >2.00 x ULN (upper limit of normal), AST, ALT > 2.5 x ULN or ALP >2.50 x ULN (upper limit of normal).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Time to progression is from the start of Docetaxel to disease progression. Patients who have not progressed at the time of study completion or who are lost to follow-up are censored at the last Vitamin D administration date. | 1 year

SECONDARY OUTCOMES:
Overall survival is defined as the time from start of Docetaxel to death due to any cause. Patients for whom no death is captured on the clinical database are censored at the last date they were known to be alive. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Taher Al-Tweigeri, MD, Principal Investigator — KFSHRC; Dahish Ajarim, MD, Study Director — KFSHRC
Locations (6):
- Kuwait Cancer Center, Kuwait City, Kuwait
- Saudi Arabia (4):
  - King Faisal Specialist Hospital & Research Center, Riyadh, Central
  - King Abdulaziz Hospital and Oncology Center, Jeddah
  - King Abdulaziz Medical City, Riyadh
  - King Fahad Medical City, Riyadh
- Tawam Hospital, Al Ain City, United Arab Emirates